CLINICAL TRIAL: NCT01779531
Title: A Phase III，Randomized ，Multi-center Clinical Trail to Compare the Outcomes of XT and XEC Adjuvant Chemotherapy Protocol in HER-negative Luminal B Breast Cancer Patients Who Reached Pathologic Response After XT Neoadjuvant Chemotherapy
Brief Title: Compare the Outcomes of XT and XEC Adjuvant Chemotherapy in HER2-negative Luminal B Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Academy of Medical Sciences (Other)
Collaborators: Chinese Anti-Cancer Association (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Liao Ning, MD,PhD, Guangdong Academy of Medical Sciences
Other Study IDs: GGHBCRG
Record Dates: First submitted 2013-01-24; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: HER2-negative Luminal B breast cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue，whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pCR，XT

SUMMARY:
Human epidermalgrowth factor receptor-2(HER2) negative Luminal B subtype breast cancer patients are included. After 4 cycles of Capecitabine combined with Docetaxel(XT) protocol neoadjuvant chemotherapy ,those who reach partial response(PR) but not pathological complete response(pCR) are randomly divided into the group treated with XT protocol and the group with Capecitabine combined with Epirubicin and Cyclophosphamide(XEC) protocol ,then compare the disease free survival(DFS) and overall survival(OS) of two subgroup.

DETAILED DESCRIPTION:
Individualized treatment of breast cancer has become one of the main directions in the clinical and research areas of breast cancer,and the individualized treatment of the estrogen receptor(ER) positive patients which covered 65% of total cases is of vital importance. Historical research showed that among the ER-positive and HER2-negative breast cancer,Luminal B breast cancer with Ki67>14% is more likely to be benefited from chemotherapy,compared with the Luminal A breast cancer with Ki67<14%. And the results of our previous research showed that, the neoadjuvant XT protocol has more than 17% pCR rate in Luminal B subtype breast cancer.However,to those who didn't reach pCR,we've got no evidence whether switching to Anthracycline-based post operative protocol can benefit them.So that,we sketch out a randomized controlled multicentric phase III clinical trail.HER2 negative Luminal B subtype breast cancer patients are included. After 4 cycles of XT protocol neoadjuvant chemotherapy ,those who reach PR but not pCR are randomly divided into the group treated with XT protocol and the group with XEC protocol ,then compare the DFS and OS of two subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Chinese population surgery patients with invasive breast cancer；
* Stage II-III；
* ER positive；
* HER2 negative；
* Ki67≥14%；
* Aged between 18 and 70 years old；
* The maximum diameter of the primary tumor greater than 1cm；
* ECOG score 0-1 points； -Have adequate baseline bone marrow and organ function reserve : absolute neutrophil count ≥ 1500/mm3, platelet count ≥ 8g/dl; the ≥ 100000/mm3 hemoglobin concentration and serum creatinine ≤ 1.5 times the upper limit of normal ; aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal , bilirubin ≤ 1.5 times the upper limit of normal ; left ventricular ejection fraction ( LVEF ) ≥ 50%

Exclusion Criteria: - Non - Chinese population of patients；

* Non- invasive cancer patients;
* Inflammatory Breast Cancer patients;
* Metastatic breast cancer patients;
* HER2 positive patients;
* Ki67<14% patients;
* No adequateBaseline bone marrow or organ function reserve;
* ECOG PS score ≥ 2 points;
* Younger than 18 years of age or greater than 70 years old;
* Already accepted therapy including chemotherapy , endocrine therapy or targeted therapy before neoadjuvant treatment;
* HER2-positive patients with left ventricular ejection fraction less than 55 % can not receiving Herceptin;
* Known allergy of docetaxel , capecitabine , epirubicin , ring phosphonamide .

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 negative Luminal B subtype breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival after adjuvant chemotherapy within five years | Within 5 years after adjuvant chemotherapy
  Within 5 years after adjuvant chemotherapy,we should evaluate disease free survival and overall survival rates as the most important outcome measure.
Overall survival after adjuvant chemotherapy within five years | Within five years after adjuvant chemotherapy
  Within 5 years after adjuvant chemotherapy,we should evaluate overall survival (OR)rates as the most important outcome measure.

SECONDARY OUTCOMES:
Imaging evaluation after neoadjuvant chemotherapy | within the 21 days after neoadjuvant chemotherapy
  After neoadjuvant chemotherapy,we should evaluate the status of patients as progress disease and then use the imaging evaluations as the proofs to plan their next therapeutic schedule or different grouping methods.

OTHER OUTCOMES:
Baseline evaluation | before the neoadjuvant chemotherapy
  Baseline evaluation includes the issues of ECOG PS scores, primary tumor Imaging evaluation, evaluation and reserve of bone marrow and organ function evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Ning, MD,PhD, Study Director — Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China